CLINICAL TRIAL: NCT00379847
Title: A 4-day, Open-Label, Multicenter Phase 3b Study of IV YM087 in Patients With Euvolemic or Hypervolemic Hyponatremia
Brief Title: An Open-Label Study of YM087 (Conivaptan) in Patients With Euvolemic or Hypervolemic Hyponatremia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cumberland Pharmaceuticals (Industry)
Responsible Party: Sr Manager Clinical Trial Registry, Astellas Pharma US, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 087-CL-080
Record Dates: First submitted 2006-09-21; First posted 2006-09-25 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-04

CONDITIONS: Hyponatremia
Keywords: hyponatremia; hypervolemic; euvolemic; treatment outcomes; YM087
MeSH Terms: conditions — Hyponatremia | interventions — conivaptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Lower dose
  Interventions: Drug: conivaptan
- 2 (Experimental): Higher dose
  Interventions: Drug: conivaptan

INTERVENTIONS:
Drug: conivaptan — IV
  Other Names: Vaprisol; YM087

SUMMARY:
This study will investigate the application of a vasopressin antagonist in the treatment of hyponatremia most likely caused by inappropriate AVP secretion. The population studied will include patients with euvolemic or hypervolemic hyponatremia.

ELIGIBILITY:
Inclusion Criteria:

* Serum sodium levels less than or equal 130mEq/L
* Euvolemic or Hypervolemic hyponatremia

Exclusion Criteria:

* Clinical evidence of volume depletion or dehydration
* Untreated severe hypothyroidism, hyperthyroidism, or adrenal insufficiency
* Uncontrolled brady-or tachyarrhythmias requiring pacemaker placement or treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2004-02; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Baseline-adjusted change in AUC for serum sodium | 96 Hours

SECONDARY OUTCOMES:
Comparison of safety between patients in each study arm | 96 Hours

CONTACTS AND LOCATIONS:
Overall Officials: Art Wheeler, MD, Study Director — Cumberland Pharmaceuticals, Inc.
Locations (28):
- United States (7):
  - Tuscon, Arizona
  - Denver, Colorado
  - Washington D.C., District of Columbia
  - Augusta, Georgia
  - Petoskey, Michigan
  - Cincinnati, Ohio
  - Columbia, South Carolina
- Israel (11):
  - Afula
  - Ashkelon
  - Hadera
  - 2 Sites, Haifa
  - Holon
  - 2 Sites, Jerusalem
  - Nahariya
  - Rehovot
  - 2 Sites, Safed
  - Tel Aviv
  - Ẕerifin
- South Africa (10):
  - Amanzimototi
  - Bellville
  - Bloemfontein
  - 2 Sites, Durban
  - 4 Sites, Johannesburg
  - Krugersdorp
  - Lyttelton
  - Pretoria
  - Somerset West
  - Soweto